CLINICAL TRIAL: NCT04900233
Title: Effect of Covid-19 Pandemic in Non Covid-19 Patients at the Emergency Surgical Department, During the Severe Restriction Phase of Lockdown in Buenos Aires. A Cohort Study.
Brief Title: Effect of Covid-19 Pandemic in Non Covid-19 Patients at the Emergency Surgical Department
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, CECILIA DANIELA JORGE, Medical doctor, Hospital Italiano de Buenos Aires
Other Study IDs: 5684
Record Dates: First submitted 2021-05-15; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Emergencies; Appendicitis; Surgical Procedure, Unspecified
MeSH Terms: conditions — COVID-19; Emergencies; Appendicitis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- Control group
  Interventions: Other: surgery
- Pandemic group
  Interventions: Other: surgery

INTERVENTIONS:
Other: surgery — emergency surgery

SUMMARY:
Introduction Most countries imposed mandatory lockdowns that were rapidly lifted, however Argentina holds the record for one of the longest quarantines in the world. General surgery emergency conditions and trauma cases still require immediate evaluation and timely resolution. The primary objective of this study was to analyze the variations in the consults, surgical outcomes and severity of disease in admissions at our department of general surgery and to study the consequences of the lockdown effect in our community.

Materials and methods An observational, ambispective study was carried out on a prospective cohort of patients who consulted with on-call surgical pathology and required hospitalization in the period from March 13th, 2020 until July 31, 2020 (PG) were included, analyzed and compared with the same period of 2019 (CG).

DETAILED DESCRIPTION:
Participation in the study does not represent any additional risk for the included participants since participation in the protocol does not include any experimental intervention and the medical care and treatment of all participants that require it will be carried out according to the current guidelines. The protocol does not contemplate any procedure or study additional to the usual care of the patient.

ELIGIBILITY:
Inclusion Criteria:

* all non-Covid-19 patients over 18 years who consulted at the emergency surgical department of Hospital Italiano de Buenos Aires and required hospitalization in the period from March 13th, 2020 until July 31, 2020 (Pandemic Group-PG) and compared with the same period of 2019 (Control Group-CG).

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: -patients over 18 years
Sampling Method: Non-Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Number of patients admitted to the emergency department | 2019-2020
  Variations in the consults the emergency department of general surgery.
Clinical presentation of the patients at the time of admission | 2019-2020
  Surgical outcomes and severity of disease in admissions at the department of general surgery.
Has the COVID-19 pandemic made a significant change in the hospital admissions? | 2019-2020
  Study the consequences of the severe restriction phase of the pandemic in the community.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No